CLINICAL TRIAL: NCT00005029
Title: Phase II Evaluation of Three-Day Topotecan (NSC 609699) in Recurrent Platinum-Sensitive Ovarian or Primary Peritoneal Cancer
Brief Title: Topotecan in Treating Patients With Recurrent Ovarian Epithelial or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067550; GOG-0146K
Record Dates: First submitted 2000-04-06; First posted 2004-07-19 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Topotecan

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of topotecan in treating patients who have recurrent ovarian epithelial or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of topotecan in patients with recurrent platinum sensitive ovarian epithelial or primary peritoneal cancer. II. Determine the nature and degree of toxicity of this treatment regimen in these patients.

OUTLINE: Patients receive topotecan IV over 30 minutes on days 1-3. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent ovarian epithelial or primary peritoneal carcinoma Bidimensionally measurable disease (ascites and pleural effusions not considered measurable) Platinum sensitive (defined as treatment free interval following response to platinum of greater than 6 months) One prior platinum based chemotherapy regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound required

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least lower limit of normal Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT and alkaline phosphatase no greater that 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No active infection requiring antibiotics No neuropathy greater than grade 1 Not pregnant Negative pregnancy test Fertile patients must use effective contraception No prior malignancy within past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic or immunologic agents Chemotherapy: See Disease Characteristics Recovered from prior chemotherapy Patients with no prior paclitaxel therapy may receive second regimen that includes paclitaxel No other prior or concurrent cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimens No prior topotecan Endocrine therapy: At least one week since prior hormonal therapy for malignant tumor Prior and concurrent hormone replacement therapy allowed Radiotherapy: No prior or concurrent radiotherapy to target sites No prior radiotherapy to greater than 25% of bone marrow Recovered from prior radiotherapy Surgery: Recovered from prior surgery Other: No prior cancer treatment that contraindicates study

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center
Locations (74):
- United States (73):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brookview Research, Inc., Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada

REFERENCES:
- [Result] Miller DS, Blessing JA, Lentz SS, McMeekin DS. Phase II evaluation of three-day topotecan in recurrent platinum-sensitive ovarian carcinoma: a gynecologic oncology group study. Cancer. 2003 Oct 15;98(8):1664-9. doi: 10.1002/cncr.11690. PMID 14534883